# Rapid Blood Culture Identification Panel in Pediatric Patients in Guatemala NCT05314816

Statistical Analysis Plan

v. 2/23/2023

#### **Statistical Analysis Plan**

Objective: to evaluate the clinical impact of the BioFire BCID2 panel in children with bacteremia in Guatemala.

<u>Study Design:</u> Pragmatic clinical trial comparing intervention to two different control groups. Intervention and concurrent control group allocated by time of blood culture positivity. Also comparing to historical controls.

<u>Primary outcome</u>: time to optimal antimicrobial therapy

#### Secondary outcomes:

- Time to effective antimicrobial therapy
- Time to pathogen identification
- Mortality
- Length of hospital stay
- Antibiotic days of therapy (DOT)
- Number of unique antibiotics
- Total ICU days

# Definitions to consider:

# **Patient Group**

Intervention= patient was enrolled in the intervention group and received the BCID2 intervention within 12h timeframe

<u>Concurrent control=</u> patient was enrolled in the study and did not receive the BCID2 intervention within 12h from blood culture positivity

- Weekday controls= Patient with positive blood culture from 1pm-11:59pm Mon-Thurs
- Weekend controls= Patient with positive blood culture from 1pm Fri- 11:59pm Sunday

<u>Per protocol</u> =patient received intervention based on original allocation.

- <u>Per protocol intervention=</u> Patient allocated to intervention based on timing of blood culture AND BCID2 was performed within 8h timeframe.
- Per protocol control= Patient allocated to control group based on timing of blood culture AND no BCID2 was performed.

<u>Protocol deviation</u>=Patient intended to remain in the allocated group, but there was an unintentional deviation from protocol.

- Protocol deviation intervention= BCID2 run between 8-12h in patient allocated to intervention.
- <u>Protocol deviation control=</u> BCID2 was sent clinically >12h from positive culture in patient allocated to control group OR patient originally allocated to intervention group but BCID2 was not performed.

#### **Sub-groups**

On-panel true pathogens = Pathogens on the BCID2 panel that are always considered real pathogens per protocol. These include, *E. faecalis, E. faecium, Listeria, Staph aureus, Strep pneumonia, Strep agalactiae, Strep pyogenes, Acinetobacter baumannii, B. fragilis, Enterobacterales, Enterobacter cloacae, E. coli, Klebsiella aerogenes, Klebsiella oxytoca, Klebsiella pneumoniae, Proteus, Salmonella, Serratia matcescens, Haemophilus influenza, Neisseria meningitidis, Pseudomonas aeruginosa, Stenotrophomonas maltophilia, Cryptococcus, Candida species.* 

<u>Gram negative on-panel pathogen</u>= On-panel true pathogens as above that are Gram negatives only. These include *Acinetobacter baumannii, B. fragilis, Enterobacterales, Enterobacter cloacae, E. coli, Klebsiella aerogenes, Klebsiella oxytoca, Klebsiella pneumoniae, Proteus, Salmonella, Serratia matcescens, Haemophilus influenza, Neisseria meningitidis, Pseudomonas aeruginosa, Stenotrophomonas maltophilia.* 

<u>Gram negative pathogen=</u> On or off-panel pathogens that are Gram negatives.

<u>On-panel classic contaminant=</u> Gram positive pathogens on the BCID2 panel that are often considered contaminants (note, may be considered real in the analysis). These include, *Staph epi, Staph lugdunensis, other Staph species, other Strep species.* 

Off-panel non-Gram negatives (other) = typically contaminants.

True pathogens (on and off panel)= excluding common contaminants.

<u>Polymicrobial</u> = More than one organism was detected by BICD2 and/or Vitek.

# Primary outcomes

Optimal antibiotic=typically narrowest spectrum agent based on predefined consensus guidelines

<u>Effective antibiotic</u>= any antibiotic susceptible based on susceptibilities even if overly broad.

<u>Time to optimal antimicrobial therapy=</u>time blood culture received in lab to time of first dose of "optimal" antibiotic. Censor at 14 days. Censor for death if "never reached" optimal. Stoppage of antibiotics if deemed a contaminant.

<u>Time to effective antimicrobial therapy</u>= time of blood culture received in lab to time of first dose of "effective" antibiotic. Censor at 14 days. Censor for death if "never reached" effective. Stoppage of antibiotics if deemed a contaminant.

<u>Clinician discretion (Intention to treat analysis (ITT))</u>=effective and optimal therapy determined based on whether **treating physicians** considered the pathogen real or a contaminant. Optimal therapy allowed additional antibiotics if the treating team was also treating for other syndromic diagnoses, such as culture-negative sepsis (if pathogen detected deemed to be a contaminant), nosocomial pneumonia, etc. if called out in diagnoses. Definitions created for optimal therapy for nosocomial pneumonia, culture-negative sepsis, etc.

- Time to effective therapy in ITT:
  - o Time from blood culture received in lab (time 0) to effective therapy
  - Time from blood culture positivity (time 0) to effective therapy
- Time to optimal therapy in ITT:
  - o Time from blood culture received in lab (time 0) to effective therapy
  - Time from blood culture positivity (time 0) to effective therapy

<u>Pathogen directed (Per protocol analysis)</u> =effective and optimal therapy based on **strict definitions** for real pathogen or contaminant created by study team. Strict optimal antibiotic definitions without allowing for additional antibiotics for culture-negative sepsis or nosocomial pneumonia, etc. Does allow for additional antibiotics for clear other indications (pyelonephritis, CAP, dacrocystitis, intra-abdominal abscess, etc.) or another organism isolated (excluding urine and trach cultures). Not allowing for more controversial diagnoses such as sepsis or nosocomial pneumonia.

- Time to effective therapy in per protocol:
  - o Time from blood culture received in lab (time 0) to effective therapy
  - o Time from blood culture positivity (time 0) to effective therapy
- Time to optimal therapy in per protocol:
  - o Time from blood culture received in lab (time 0) to effective therapy
  - o Time from blood culture positivity (time 0) to effective therapy

#### **Secondary outcomes**

<u>Time to pathogen identification=</u> Time from time of blood culture receipt in lab (time 0) to identification of a pathogen. For control patients, this is the time to Vitek. For intervention patients, this is the time to BCID2 was positive for an on-panel pathogen or time to vitek if the BCID2 was negative.

- Control: time to Vitek
- Intervention:
  - If BCID2 positive → calculate time to BCID2 result
  - If BCID2 negative → calculate time to Vitek

<u>Total antibiotic days=</u>all days that patient was on antibiotics (any dose of antibiotic) from date that blood culture was drawn. Capped at 14 days or date of death.

Antibiotic days of therapy = Sum of antibiotics each day over 14-day period. For example if 2 antibiotics were each given over 5 days, this would count as 10 DOT.

Number of different antibiotics=Number of unique antibiotics given over the 14-day period.

Length of stay=date admitted to date patient left the study (date of death/discharge or lapse of 30 days). Censor at 30 days.

<u>Total ICU days=</u>date admitted in ICU to date transferred out or date of death/discharge. Censor at 30 days.

<u>Time to death=</u> Time from blood culture obtained to time of death.

Number of deaths within 24h of blood culture draw= Use time of death calculation above to determine the number of patients who died <24h

#### Overview of Analyses to perform:

- All interventions vs. all concurrent controls (including protocol deviations) vs. historical controls
  - Demographics
  - o All outcomes (primary and all secondary endpoints)
  - o Sensitivity analysis comparing weekday vs. weekend controls
- Per protocol controls vs. per protocol intervention (excluding protocol deviations)
  - o Demographics
  - o All outcomes (primary and all secondary endpoints)
- Clinician discretion (ITT) analysis (controls vs. interventions)

- o Number of contaminants vs. true pathogens
- Time to optimal therapy
- Time to effective therapy
- Pathogen directed (Per protocol) analysis (controls vs. interventions)
  - o Number of contaminants vs. true pathogens
  - o Time to optimal therapy
  - Time to effective therapy
- Gram negatives only (on- and off- panel)
  - o Demographics
  - Time to optimal therapy
  - Time to effective therapy
  - Mortality
- On-panel true pathogens only
  - o Demographics
  - o Time to optimal therapy
  - Time to effective therapy
  - Mortality
- On-panel Gram negatives only
  - o Demographics
  - Time to optimal therapy
  - Time to effective therapy
  - Mortality
- True pathogens (on and off panel)
  - o Demographics
  - o Time to optimal therapy
  - o Time to effective therapy
  - Mortality

Figure 1: CONSORT Diagram

**Table 1: Patient Characteristics** 

| | All<br>Intervention<br>N = 135 | All Concurrent Control N = 219 | p-value<br>(interv. vs.<br>concurrent<br>control) | Weekend<br>controls<br>N=XX | p-value<br>(interv.<br>Vs.<br>weekend) | Weekday<br>controls<br>N=XX | p-value<br>(interv.<br>Vs.<br>weekday) | Historical<br>controls<br>N=99 | p-value<br>(intervention<br>vs. historical<br>control) |
|---|---|---|---|---|---|---|---|---|---|
| Age in months (median, IQR)* | | | | | , | | ,, | | |
| Categorical age<br>groups (0-30 days, 1-<br>5.99mo, 6-11.99mo,<br>12month-<br>23.99month, 24<br>month-4.99y, >=5y)** | | | | | | | | | |
| Female (n, %)** | | | | | | | | | |
| No antecedent medical conditions (N, %)** | | | | | | | | | |
| Immunocompromised (N, %)** | | | | | | | | | |
| Central line (N, %)** | | | | | | | | | |
| Required ICU stay (N, %)** | | | | | | | | | |

<sup>\*</sup>Wilcoxon test of medians

Table 1A: Supplemental table with demographics from sub-groups.

| Per p | orotocol Pe | er p- | True on- | True on- | p- | All | All GN | p- | All GN | p-value | On- | On- | p- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Inter | vention prot | cocol value | panel | panel | value | Gram | control | value | weekDAY | (compare | panel | panel | value |
| | Con | itrol | pathogen | Pathogen | | negative | | | controls | to GN | GN | GN | |
| | | | Intervention | controls | | (GN) | | | | interv.) | Interv. | control | |
| | | | | | | Interv. | | | | | | | |

<sup>\*\*</sup>chi-square test

| Age in months (median, IQR)* |
|---|
| Categorical age<br>groups (0-30 days, 1-<br>5.99mo, 6-11.99mo,<br>12month-<br>23.99month, 24<br>month-4.99y, >=5y)** |
| Female (n, %)** |
| No antecedent medical conditions (N, %)** |
| Immunocompromised (N, %)** |
| Central line (N, %)** |
| Required ICU stay (N, %)** |

Table 2: Organisms isolated in culture (Vitek)

| ORGANISM | INTERVENTION<br>N=135 (%)* | CONCURRENT<br>CONTROL<br>N=219 (%)* | STUDY TOTAL<br>N=354 (%)* | HISTORICAL<br>CONTROLS<br>N=99 (%)* | Weekend<br>controls<br>N=XX (%) | Weekday<br>controls<br>N=XX (%) |
|---|---|---|---|---|---|---|
| BCID2 Panel organisms | | | | | | |
| Acinetobacter calcoacetius-baumannii complex (n, %) | | | | | | |
| Bacteroides fragilis | | | | | | |
| Haemophilus influenzae<br>Neisseria meningitidis | | | | | | |
| Pseudomonas aeruginosa | | | | | | |
| Stenotrophomonas<br>maltophilia | | | | | | |

| Escherichia coli Escherichia coli Klebsiella aerogenes Klebsiella pneumoniae group Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecalis Estaphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pyogenes (Group A) Candida albicans Candida krusei Candida tropicalis Cryptococcus Candida tropicalis Candida tropicalis Candida tropicalis Candida tropicalis Cryptococcus | Enterobacter cloacae |
|---|---|
| Escherichia coli Iklebsiella aerogenes Iklebsiella oxytoca Iklebsiella oxytoca Iklebsiella preumoniae group Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus aglactiae (Group B) Streptococcus pyogenes (Group A) Candida albicans Candida glabrata Candida glabrata Candida trusei Candida trusei Candida tropicalis Candida tropicalis Candida proposiosis Candida tropicalis Cryptococcus | |
| Klebsiella progenes Klebsiella protroca Klebsiella protroca Klebsiella protroca Klebsiella protroca Klebsiella protroca Brotroca Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecalis Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Staphylococcus (Group B) Streptococcus agalactiae (Group B) Streptococcus protrococcus protrococ | |
| Klebsiella oxytoca Klebsiella pneumoniae group Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecilis Enterococcus faecilim Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pneumoniae Streptococcus Candida albicans Candida glabrata Candida glabrata Candida grapsilosis Candida tropicalis Candida tropicalis Candida tropicalis Candida tropicalis Candida tropicalis Cryptococcus | |
| Klebsiella pneumoniae group Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidernidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pogenes Streptococcus pogenes Candida aluris Candida krusei Candida trusei | |
| group Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida krusei Candida tropicalis Candida tropicalis Candida tropicalis Candida tropicalis Candida tropicalis Cryptococcus Cardida tropicalis Candida tropicalis Candida tropicalis Cryptococcus | |
| Proteus spp. Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus aureus Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida fauris Candida parapsilosis Candida tropicalis Cryptococcus | - |
| Salmonella spp. Serratia marcescens Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida glabrata Candida parapsilosis Candida tropicallis Candida tropicallis Cryptococcus Conyptococcus Conyptoccus Cony | |
| Serratia marcescens Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida prapsilosis Candida tropicalis Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus | |
| Enterococcus faecalis Enterococcus faecium Listeria monocytogenes Staphylococcus aureus Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida glabrata Candida grapsilosis Candida tropicalis Candida tropicalis Cryptococcus Cryptococcus Compocus poole (Group A) Candida tropicalis Candida tropicalis Cryptococcus Cryptococcus | |
| Enterococcus faecium Listeria monocytogenes Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida glabrata Candida parapsilosis Candida tropicalis Cryptococcus Cryptococcus Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus Candida tropicalis Candida tropicalis Candida tropicalis Cryptococcus | |
| Listeria monocytogenes Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida glabrata Candida parapsilosis Candida tropicalis Cryptococcus Cryptococcus Companis Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus Candida canres Candida tropicalis Cryptococcus Candida tropicalis Cryptococcus | |
| Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida glabrata Candida glabrata Candida brusei Candida tropicalis Candida tropicalis Cryptococcus Cryptococcus | |
| Staphylococcus epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | |
| epidermidis Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida tropicalis Cryptococcus Cryptococcus | |
| Staphylococcus lugdunensis Streptococcus agalactiae (Group B) Streptococcus proeumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | |
| Iugdunensis Streptococcus agalactiae (Group B) Streptococcus Streptococcus pneumoniae Streptococcus pyogenes (Group A) Streptococcus pyogenes (Group A) Streptococcus Candida albicans Streptococcus Candida glabrata Streptococcus Candida parapsilosis Streptococcus Candida tropicalis Streptococcus | |
| Streptococcus agalactiae (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida parapsilosis Candida prapsilosis Candida tropicalis Cryptococcus | |
| (Group B) Streptococcus pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Candida tropicalis Cryptococcus Cryptococcus | |
| Streptococcus progenes Streptococcus progenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | |
| pneumoniae Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | |
| Streptococcus pyogenes (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | Streptococcus |
| (Group A) Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | pneumoniae |
| Candida albicans Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | Streptococcus pyogenes |
| Candida auris Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | |
| Candida glabrata Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | Candida albicans |
| Candida krusei Candida parapsilosis Candida tropicalis Cryptococcus | Candida auris |
| Candida parapsilosis Candida tropicalis Cryptococcus | Candida glabrata |
| Candida tropicalis Cryptococcus | |
| Candida tropicalis Cryptococcus | Candida parapsilosis |
| Cryptococcus | |
| | neoformans/gattii |

| Other coagulase-negative |
|----------------------------|
| Staphylococcus species |
| Other Streptococcus |
| species |
| Total on-panel targets |
| Non-BCID2 organisms |
| Bacillus species |
| Achromobacter species |
| Burkholderia species |
| Shewanella species |
| Sphingomonas species |
| Other Acinetobacter |
| species |
| Pantoea species |
| Other Pseudomonas |
| species |
| Alloiococcus species |
| Aeromonas species |
| Leuconostoc species |
| Kocuria species |
| Citrobacter freundii |
| Gram positive Bacillus (no |
| ID) |
| Moraxella species |
| Pandoraea species |
| Kluyvera species |
| Total non-BCID2 targets |

<sup>\*</sup>n= number of cultures. Some cultures grew more than one isolate. Percentage of each organism was calculated from the total number of cultures.

Table 2A: Supplemental table of organisms for sub-groups. (Will likely add historical controls to supplemental table)

| ORGANISM | Per protocol<br>Intervention<br>N=112 (%)* | Per protocol<br>controls<br>N=192 (%)* | Protocol deviation interventions N=23 (%)* | Protocol<br>deviation<br>controls<br>N=27(%)* |
|---|---|---|---|---|
| BCID2 Panel organisms | | | | |
| Acinetobacter calcoacetius-baumannii complex Bacteroides fragilis | | | | |
| Haemophilus influenzae | | | | |
| Neisseria meningitidis Pseudomonas aeruginosa | | | | |
| Stenotrophomonas<br>maltophilia | | | | |
| Enterobacter cloacae complex | | | | |
| Escherichia coli | | | | |
| Klebsiella aerogenes | | | | |
| Klebsiella oxytoca | | | | |
| Klebsiella pneumoniae<br>group | | | | |
| Proteus spp. | | | | |
| Salmonella spp. | | | | |
| Serratia marcescens | | | | |
| Enterococcus faecalis | | | | |
| Enterococcus faecium | | | | |
| Listeria monocytogenes | | | | |
| Staphylococcus aureus | | | | |
| Staphylococcus<br>epidermidis | | | | |
| Staphylococcus<br>lugdunensis | | | | |

| Chua ata aa aa u a a aala ati a a |
|-----------------------------------|
| Streptococcus agalactiae |
| (Group B) |
| Streptococcus |
| pneumoniae |
| Streptococcus pyogenes |
| (Group A) |
| Candida albicans |
| Candida auris |
| Candida glabrata |
| Candida krusei |
| Candida parapsilosis |
| Candida tropicalis |
| Cryptococcus |
| neoformans/gattii |
| Other coagulase-negative |
| Staphylococcus species |
| Other Streptococcus |
| species |
| Total on-panel targets |
| Non-BCID2 organisms |
| Bacillus species |
| Achromobacter species |
| Burkholderia species |
| Shewanella species |
| Sphingomonas species |
| Other Acinetobacter |
| species |
| Pantoea species |
| Other Pseudomonas |
| species |
| Alloiococcus species |
| Aeromonas species |
| Leuconostoc species |

| Kocuria species |
|----------------------------|
| Citrobacter freundii |
| Gram positive Bacillus (no |
| ID) |
| Moraxella species |
| Pandoraea species |
| Kluyvera species |
| Total non-BCID2 targets |

## **Table 3: Outcomes**

| | Interventions<br>N=135 | Concurrent<br>Controls<br>N=219 | p-value | Weekend<br>control | p-value<br>(interv.<br>vs.<br>weekend) | Weekday<br>control | p-value<br>(interv.<br>vs.<br>weekday) | Historical<br>controls<br>N=99 | p-value<br>(interven.<br>vs.<br>historic) |
|---|---|---|---|---|---|---|---|---|---|
| Median time to optimal therapy per protocol (XX | | | | | , | | | | , |
| hours) | | | | | | | | | |
| Median time to effective therapy per protocol (XX hours) | | | | | | | | | |
| Median time to pathogen identification (XX hours) | | | | | | | | | |
| All-cause mortality (n, %) | | | | | | | | | |
| Median time<br>to death from | | | | | | | | | |

| blood culture | | |
|-----------------|------|------|
| obtained (XX | | |
| days) | | |
| Deaths within | | |
| 24h of blood | | |
| culture drawn | | |
| (N, %)** | | |
| Deaths from | | |
| sepsis (N, %) | | |
| Deaths from | | |
| other causes | | |
| (N, %) | | |
| Cause of death | | |
| unknown (N, %) | | |
| Median LOS (XX | | |
| days) | | |
| Median ICU | | |
| days (XX days) | | |
| Median total | | |
| antibiotic days | | |
| (XX days) | | |
| Median | | |
| antibiotics DOT | | |
| Number of | <br> | <br> |
| unique | | |
| antibiotics in | | |
| 14-day period | | |
| 14 day period | | |

# Table 3A: For NICU kids only

| Int | terventions | Concurrent | p-value | Weekend | p-value | Weekday | p-value | Historical | p-value |
|---|---|---|---|---|---|---|---|---|---|
| N= | =135 | Controls | | control | | control | | controls | |
| | | N=219 | | | | | | N=99 | |

| optimal therapy (XX hours) Median time to effective therapy (XX hours) Median time to pathogen identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from ode to the third of the thir | | | ı | ı | T |
|---|---|---|---|---|---|
| (XX hours) Median time to effective therapy (XX hours) Median time to pathogen identification (XX hours) All-cause mortality (n, %) Median time to to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (n, %)** Deaths from sepsis (n, %) Deaths from sepsis (n, %) Deaths from other causes (n, %) Median LOS (XX days) | Median time to | | | | |
| Median time to effective therapy (XX hours) Median time to pathogen identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (n, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median LOS (XX days) | | | | | |
| effective therapy (XX hours) Median time to pathogen identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median LOS (XX days) Median ICU | | | | | |
| therapy (XX hours) Median time to pathogen identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (n, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | Median time to | | | | |
| Nedian time to pathogen | effective | | | | |
| Median time to pathogen identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | therapy (XX | | | | |
| pathogen identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (n, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | hours) | | | | |
| identification (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | Median time to | | | | |
| (XX hours) All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | pathogen | | | | |
| All-cause mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | identification | | | | |
| mortality (n, %) Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | (XX hours) | | | | |
| Median time to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | All-cause | | | | |
| to death from blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | mortality (n, %) | | | | |
| blood culture obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | Median time | | | | |
| obtained (XX days) Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | to death from | | | | |
| Deaths within 24h of blood | blood culture | | | | |
| Deaths within 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | obtained (XX | | | | |
| 24h of blood culture drawn (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | days) | | | | |
| culture drawn (N, %)** Deaths from sepsis (N, %) Sepsis (N, %) Deaths from other causes (N, %) Sepsis (N, %) Cause of death unknown (N, %) Sepsis (N, %) Median LOS (XX days) Sepsis (N, %) | Deaths within | | | | |
| (N, %)** Deaths from sepsis (N, %) Deaths from other causes (N, %) 0 Cause of death unknown (N, %) 0 Median LOS (XX days) 0 Median ICU 0 | 24h of blood | | | | |
| Deaths from sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | culture drawn | | | | |
| sepsis (N, %) Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | (N, %)** | | | | |
| Deaths from other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | Deaths from | | | | |
| other causes (N, %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | sepsis (N, %) | | | | |
| %) Cause of death unknown (N, %) Median LOS (XX days) Median ICU | Deaths from | | | | |
| Cause of death unknown (N, %) Median LOS (XX days) Median ICU | other causes (N, | | | | |
| unknown (N, %) Median LOS (XX days) Median ICU | %) | | | | |
| Median LOS (XX days) Median ICU | Cause of death | | | | |
| days) Median ICU | unknown (N, %) | <br> | | | |
| Median ICU | Median LOS (XX | | | | <br> |
| | days) | | | | |
| days (XX days) | Median ICU | | | | |
| | days (XX days) | | | | |

| Median total<br>antibiotic days |
|---------------------------------|
| (XX days) |
| Median |
| antibiotics DOT |
| Number of |
| unique |
| antibiotics in |
| 14-day period |

Table 3B: For non-NICU patients only

| | Interventions<br>N=135 | Concurrent<br>Controls<br>N=219 | p-value | Weekend<br>control | p-value | Weekday<br>control | p-value | Historical controls N=99 | p-value |
|---|---|---|---|---|---|---|---|---|---|
| Median time to optimal therapy | | | | | | | | | |
| (XX hours) | | | | | | | | | |
| Median time to | | | | | | | | | |
| effective | | | | | | | | | |
| therapy (XX | | | | | | | | | |
| hours) | | | | | | | | | |
| Median time to | | | | | | | | | |
| pathogen | | | | | | | | | |
| identification | | | | | | | | | |
| (XX hours) | | | | | | | | | |
| All-cause | | | | | | | | | |
| mortality (n, %) | | | | | | | | | |
| Median time | | | | | | | | | |
| to death from | | | | | | | | | |
| blood culture | | | | | | | | | |
| obtained (XX | | | | | | | | | |
| days) | | | | | | | | | |

| Deaths within |
|------------------|
| 24h of blood |
| culture drawn |
| (N, %)** |
| Deaths from |
| sepsis (N, %) |
| Deaths from |
| other causes (N, |
| %) |
| Cause of death |
| unknown (N, %) |
| Median LOS (XX |
| days) |
| Median ICU |
| days (XX days) |
| Median total |
| antibiotic days |
| (XX days) |
| Median |
| antibiotics DOT |
| Number of |
| unique |
| antibiotics in |
| 14-day period |

Table 3C: Table of outcomes with sub-groups for all units

| | Per | Per | p- | All Gram | All Gram | p- | All GN | p-value | True on- | True on- | р- | On-panel | On- | p-valu |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | protocol | protocol | value | negative | negative | value | weekDAY | (compar | panel | panel | value | Gram | panel | |
| | interventio | Controls | ' l | interventio | controls | | controls | e to GN | pathoge | pathogen | | neg | Gram | |
| | ns | 1 | ' l | ns | ' | | Į į | interv.) | <sup>l</sup> n j | controls | | interv | neg | |
| | | | ' l | ' | ' 1 | | ļ , | ļ , | intervent | !<br>! | | ! | control | |
| L | | | ' <u></u> | <u>'</u> | <u> </u> | | Į į | <u> </u> | ions | !<br>i | | ' <u> </u> | <u> </u> | |

| | <br> | <br> | <br> | <br> | <br> | | <br> |
|---|---|---|---|---|---|---|---|
| Median time to optimal therapy | | | | | | | |
| (XX hours) | | | | | | | |
| Median time to | | | | | | | |
| effective therapy | | | | | | | |
| (XX hours) | | | | | | | |
| Median time to | | | | | | | |
| pathogen | | | | | | | |
| identification (XX | | | | | | | |
| hours) | | | | | | | |
| All-cause | | | | | | | |
| mortality (n, %) Median time to | | | | | | | |
| death from | | | | | | | |
| blood culture | | | | | | | |
| obtained (XX | | | | | | | |
| days) | | | | | | | |
| Deaths within | | | | | | | |
| 24h of blood | | | | | | | |
| culture drawn | | | | | | | |
| (N, %)** | | | | | | | |
| Deaths from | | | | | | | |
| sepsis (N, %) | | | | | | | |
| Deaths from | | | | | | | |
| other causes (N, | | | | | | | |
| %) | | | | | | 1 | |
| Cause of death | | | | | | | |
| unknown (N, %) | | | | | | | |
| Median LOS (XX | | | | | | | |
| days) | | | | | | | |
| Median ICU days | | | | | | | |
| (XX days) | | | | | | | |

| Median total |
|--------------------|
| antibiotic days |
| (XX days) |
| Median |
| antibiotics DOT |
| Number of |
| unique |
| antibiotics in 14- |
| day period |

# Table 4: BCID2/Vitek discrepancies in intervention patients

| | Number of patients (N, %) |
|----------------------------------------------|---------------------------|
| BCID2/Vitek agreed | |
| BCID2/Vitek disagreed | |
| BCID2 positive, Vitek negative | |
| BCID2 negative, Vitek positive | |
| Species misidentification | |
| Resistance gene did not match susceptibility | |
| Organism not on panel | |

# Other parameters:

- Look at distribution (median with IQR) of time between BCID2 result and team notification (only for intervention patients).
- Look at distribution (median with IQR) of time between BCID2 execution and team notification (only for intervention patients).
- Age distribution and gender between those excluded via initial screening and those included (initially enrolled).

Figures: Kaplan Meier curves for time to optimal and time to effective therapy (using both intention to treat AND per protocol analyses)

 $\mathbf{1}^{\text{st}}$  way- time of blood culture draw as time  $\mathbf{0}$ 

2<sup>nd</sup> way- time of blood culture positivity as time 0

Figure 1: Compare interventions vs. concurrent controls vs. Historical controls (all pathogens)

Figure 1A: time to effective therapy ITT

Figure 1B: time to effective therapy per protocol

Figure 1C: time to optimal therapy ITT

Figure 1D: time to optimal therapy per protocol

Figure 1E: time to death (deaths only)

Figure 2: Compare interventions vs. concurrent controls vs. Historical controls (Gram negative rods on-panel and off-panel)

Figure 3: Compare interventions vs. concurrent controls vs. Historical controls (True on-panel pathogens only)

Figure 4: Compare interventions vs. concurrent controls vs. Historical controls (on-panel Gram negative pathogens only)